CLINICAL TRIAL: NCT06753266
Title: OPTIMIST Optimizing OR Simulation in MEDI 045 Anesthesia Program: Trends, Bias Reduction, and Strategic Improvements and Shaping Future Practices OPTIMIST
Brief Title: Optimizing OR Simulation in MEDI 045: Bias Reduction and Strategic Improvements (OPTIMIST)
Acronym: OPTIMIST
Status: Active, not recruiting | Type: Observational
Sponsor: Walid Mohamed Ragab Mohamed Badwi (Other Government)
Responsible Party: Sponsor-Investigator, Walid Mohamed Ragab Mohamed Badwi, Resident in Anesthesia, Instructor in MEDI 045, King Saud University College of Medicine., King Saud Medical City
Organization: King Saud Medical City (Other Government)
Other Study IDs: KSU-ORSim-2024
Record Dates: First submitted 2024-12-16; First posted 2024-12-31 (Actual); Last update posted 2024-12-31 (Actual); Status verified 2024-12

CONDITIONS: Competency-Based Education; Continuity of Patient Care; Medical Education
Keywords: Simulation-Based Training; Anesthesia Education; Patient Safety; Operating Room Simulation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study explores the evolving landscape of operating room (OR) simulation by identifying key trends, addressing potential biases, and providing actionable recommendations for improvement. Using data-driven analysis, the research uncovers patterns in skill development and decision-making, offering insights into the effectiveness of current OR simulation programs. The study also tackles biases in data collection, including selection and response bias, ensuring the reliability of findings.

DETAILED DESCRIPTION:
The effectiveness of simulation training is crucial in medical education, particularly for skills retention and perceived effectiveness. This section evaluates the overall effectiveness of SimMan3G sessions in enhancing clinical skills among participants.

Objectives

* To analyze the correlation between the number of SimMan3G sessions and skill retention.
* To assess the perceived effectiveness of simulation training.
* To provide actionable recommendations for improving simulation training effectiveness.

ELIGIBILITY:
Inclusion Criteria:

* Participants enrolled in the MEDI 045 anesthesia program at King Saud Medical City.
* Medical students or trainees with prior exposure to basic clinical simulation.
* Aged 18 years or older.
* Willingness to participate in simulation-based training sessions.
* Ability to provide informed consent.

Exclusion Criteria:

* Participants with prior advanced simulation training in anesthesia.
* Individuals with documented cognitive impairments or learning disabilities that may interfere with the study tasks.
* Refuse to participate in post-simulation assessments or follow-ups.
* Lack of fluency in the language of instruction used in the simulation.

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: The study population consists of medical trainees enrolled in the MEDI 045 anesthesia program at King Saud Medical City.
  Participants will include individuals with varying levels of clinical experience who are eligible for simulation-based training.
  Participants will be randomly selected from a list of eligible trainees in the MEDI 045 program.
Sampling Method: Non-Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2024-11-15 (Actual); Primary Completion 2025-01-15 (Estimated); Study Completion 2025-03-15 (Estimated)

PRIMARY OUTCOMES:
Change in Cognitive Bias in Clinical Decision-Making | Immediately after simulation training (within 1 day) Over 6 months post-training
  Evaluate the change in cognitive bias during simulated clinical scenarios using the Cognitive Bias Assessment Tool (CBAT). This tool assesses the presence of cognitive biases (e.g., confirmation bias, anchoring bias) in decision-making.
  The unit of measure will be the percentage of bias-free decisions or correct decisions made by participants, based on the CBAT scoring system.
  The assessment will occur immediately after simulation training (within 1 day) and again 6 months post-training to measure both immediate and long-term changes in cognitive bias.

CONTACTS AND LOCATIONS:
Locations (4):
- Saudi Arabia (4):
  - King Saud University MedicalCity, Riyadh, Riydh
  - King Saud University MedicalCity, Riyadh
  - King Saud University , College of Medicine, Anesthesia Department, Riyadh
  - King Saud University Medical City (KSUMC), College of Medicine, Riyadh